CLINICAL TRIAL: NCT01528813
Title: AVALIAÇÃO DO USO DO LASER ERBIUM-DOPED YTTRIUM ALUMINIUM GARNET (Er:YAG) ASSOCIADO AO ESMALTE DE AMOROLFINA NO TRATAMENTO DA ONICOMICOSE
Brief Title: Erbium-doped Yttrium Aluminium Garnet Laser(Er:Yag)Associated With Amorolfine Lacquer in the Treatment of Onychomycosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brasilia University Hospital (Other)
Responsible Party: Principal Investigator, Izelda Maria Carvalho Costa, Adjunct Professor, Brasilia University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUB-UnB OnychoLASER
Record Dates: First submitted 2012-02-05; First posted 2012-02-08 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Onychomycosis
Keywords: Erbium-doped yttrium aluminium garnet laser; Er:YAG; Amorolfine lacquer; Dermatophytes; Subungual distal lateral onychomycosis; Drug delivery
MeSH Terms: conditions — Onychomycosis | interventions — Lasers, Solid-State; amorolfine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Er:YAG + amorolfine lacquer (Active Comparator): 30 ungual units affected by onychomycosis due to dermatophytes
  Interventions: Device: Er:YAG laser + amorolfine lacquer
- Amorolfine lacquer (Placebo Comparator): 30 ungual units affected by onychomycosis due to dermatophytes
  Interventions: Drug: Amorolfine lacquer

INTERVENTIONS:
Device: Er:YAG laser + amorolfine lacquer — To each compromised ungual unit randomly assigned to this group it will be applied a single session of Er:YAG laser to the ungual lamina in the beginning of study. Onwards, amorolfine lacquer will be applied weekly for a period of 06 months.
  Other Names: Loceryl; Er:YAG laser
  Arms: Er:YAG + amorolfine lacquer
Drug: Amorolfine lacquer — To each compromised ungual unit randomly assigned to this group, it will be applied amorolfine lacquer weekly for a period of 06 months.
  Other Names: Loceryl
  Arms: Amorolfine lacquer

SUMMARY:
The study aims to investigate the effectiveness of a single application of Er:YAG laser to the nail plate in increasing the efficacy of the amorolfine lacquer used in the treatment of onychomycosis (fungal infection of nails) cause by dermatophyte molds. This clinical trial respective involve 30 subjects with hands or feet distal-lateral subungual onychomycosis (a kind of onychomycosis that does not affect the ungual matrix). The patients will receive treatment for 6 months meanwhile they will be followed up to access efficacy of the treatment by means of the clearance of nail plate infection.

DETAILED DESCRIPTION:
This is a trial study involving 30 subjects with onychomycosis of hands or feet. The patient must have at least 2 injured nails as each affected nail will receive a different treatment - self-controlled study design.

Therefore, each nail out of two from a single patient will be randomized into the following study arms:

Group A of nails - will receive only weekly application of amorolfine lacquer for a total of 6 months.

Group B of nails - will receive a single application of Er:YAG laser followed by weekly application of amorolfine lacquer for a total of 6 months.

At the end of 6 months the data from both groups, A and B, regarding *clinical cure, *mycological cure and *extent of damage to the nail plates will be analyzed using specific tests.

ELIGIBILITY:
Inclusion Criteria:

* 19-60 year-old
* preserved cognitive status
* direct mycological examination or culture showing infection of hands or feet nails by dermatophyte molds

Exclusion Criteria:

* diabetes type 1 or 2; peripheral vascular disease
* having undergone any treatment in the last 6 months
* peripheral nerve disorders (e.g. peripheral neuropathy, Hansen's disease, etc)
* willing to paint nail during the study
* high blood pressure
* use of any immunosuppressive drugs; congenital or acquired immunodeficiency

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Extent of nail plate damage | 6 months
  At the beginning and after 6 months of treatment both the group, A and B, will have the length from nail cuticle to the closest point of damage to the nail plate measured by a millimeter scale. It will later be accessed to determine the clearance rate of the nail plate achieved with each treatment

SECONDARY OUTCOMES:
Mycological cure | 6 months
  After 6 months of treatment both the group, A and B, will be accessed by direct mycological examination and culture to evaluate mycological cure
Clinical cure | 6 months
  After 6 months of treatment both the group, A and B, will be accessed by dermatological examination to evaluate clinical cure

CONTACTS AND LOCATIONS:
Overall Officials: Orlando O Morais, M.D., Principal Investigator — University of Brasilia
Locations (1):
- University Hospital of Brasilia, Brasília, Federal District, Brazil

REFERENCES:
- [Derived] Morais OO, Costa IM, Gomes CM, Shinzato DH, Ayres GM, Cardoso RM. The use of the Er:YAG 2940nm laser associated with amorolfine lacquer in the treatment of onychomycosis. An Bras Dermatol. 2013 Sep-Oct;88(5):847-9. doi: 10.1590/abd1806-4841.20131932. PMID 24173203